CLINICAL TRIAL: NCT00848380
Title: Management of Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. Dirk Schneider , Medical Affairs & Regulatory Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CCH-DUM-2008/2
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Cardiovascular Risk Factors; Cardiovascular Diseases
Keywords: Hypertension; hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hypertension and hyperlipidemia and other CV risk factors

SUMMARY:
This practical experience should report a retrospective collection of data regarding cardiovascular risk factors of cardiovascular diseases. The goal is an evaluation of the development of the risk profile of cardiovascular patients with simultaneous treatment of hypertension and hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Patients received a anti-hypertension treatment in addition to cholesterol lowering treatment during the observation period
* Patients received a cholesterol lowering treatment in addition to hypertension treatment during the observation period
* Patients received during the observation time new cholesterol lowering and hypertension treatment

Exclusion Criteria:

* Patients received during the observation time only cholesterol lowering or only anti-hypertension treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hypertension and hyperlipidemia and other CV risk factors
Sampling Method: Probability Sample
Enrollment: 1492 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The goal is an evaluation of the development of the risk profile of cardiovascular patients with simultaneous treatment of hypertension and hyperlipidemia. | Inclusion visit, 6 to 9 months before inclusion visit and / or 12 to 15 months before inclusion visit

CONTACTS AND LOCATIONS:
Locations (36):
- Switzerland (36):
  - Research Site, Frick, Canton of Aargau
  - Research Site, Neuenhof, Canton of Aargau
  - Research Site, Riehen, Canton of Basel-City
  - Research Site, Thun, Canton of Bern
  - Research Site, Wynigen, Canton of Bern
  - Research Site, Geneva, Canton of Geneva
  - Research Site, Le Lignon, Canton of Geneva
  - Research Site, Meyrin, Canton of Geneva
  - Research Site, Schwyz, Canton of Schwyz
  - Research Site, Gerlafingen, Canton of Solothurn
  - Research Site, Lohn SO, Canton of Solothurn
  - Research Site, Zuchwil, Canton of Solothurn
  - Research Site, Rorschach, Canton of St. Gallen
  - Research Site, Sankt Gallen, Canton of St. Gallen
  - Research Site, Bassins, Canton of Vaud
  - Research Site, Gland, Canton of Vaud
  - Research Site, Lausanne, Canton of Vaud
  - Research Site, Montreux, Canton of Vaud
  - Research Site, Nyon, Canton of Vaud
  - Research Site, Zug, Canton of Zug
  - Research Site, Affoltern am Albis, Canton of Zurich
  - Research Site, Feldmeilen, Canton of Zurich
  - Research Site, Herrliberg, Canton of Zurich
  - Research Site, Langnau am Albis, Canton of Zurich
  - Research Site, Richterswil, Canton of Zurich
  - Research Site, Rüti, Canton of Zurich
  - Research Site, Zurich, Canton of Zurich
  - Research Site, Arbedo, Canton Ticino
  - Research Site, Bellinzona, Canton Ticino
  - Research Site, Claro, Canton Ticino
  - Research Site, Coldrerio, Canton Ticino
  - Research Site, Locarno, Canton Ticino
  - Research Site, Lugano, Canton Ticino
  - Research Site, Muralto, Canton Ticino
  - Research Site, Andeer, Kanton Graubünden
  - Research Site, Ilanz, Kanton Graubünden